CLINICAL TRIAL: NCT03221751
Title: Prazosin and CSF Biomarkers in mTBI
Brief Title: Prazosin and Cerebrospinal Fluid (CSF) Biomarkers in Mild Traumatic Brain Injury (mTBI)
Acronym: PoND
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: staffing issues and COVID
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: B2180-P; 1I21RX002180-01 (NIH)
Record Dates: First submitted 2017-07-13; First posted 2017-07-19 (Actual); Results first posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Dementia
Keywords: randomized controlled trial
MeSH Terms: conditions — Dementia | interventions — Prazosin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prazosin (Experimental): Subjects will be titrated up to the maximum dose or the maximum tolerated dose based on a dosing algorithm. The maximum dose is 5 mg in the morning, 5 mg in the afternoon and 15 mg at bedtime.
  Interventions: Drug: prazosin hydrochloride
- Placebo (Placebo Comparator): Subjects will be titrated up to the maximum dose or the maximum tolerated dose based on a dosing algorithm. The maximum dose is 5 mg in the morning, 5 mg in the afternoon and 15 mg at bedtime.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: prazosin hydrochloride — Prazosin is an oral capsule. It is an alpha-1 antagonists.
  Other Names: Minipress
  Arms: Prazosin
Drug: placebo — Placebo is an inert oral capsule identical in appearance to prazosin capsules.
  Other Names: inactive drug; sugar pill
  Arms: Placebo

SUMMARY:
Mild traumatic brain injury (mTBI) from explosions is the "signature injury" of Veterans who have deployed to the wars in Afghanistan and Iraq. Although the immediate effects of a single mTBI usually resolve over days or weeks, multiple mTBIs can lead to both persistent symptoms and, years later, to two fatal progressive brain diseases, chronic traumatic encephalopathy (CTE) and Alzheimer's disease (AD). It is believed that CTE and AD are caused by nerve damaging chemicals called tau and beta amyloid produced by the brain but which are not removed from the brain in a normal manner in persons with mTBIs. The investigators will determine in Veterans who experienced mTBIs whether a clinically available drug called prazosin increases removal of tau and beta amyloid from the brain. This will be accomplished by seeing if prazosin reduces the amount of tau and beta amyloid in the spinal fluid that surrounds the brain. If the investigators find such reductions, prazosin will be evaluated as a preventative treatment for CTE and AD in future studies.

DETAILED DESCRIPTION:
A majority of neurodegenerative dementing disorders, including Alzheimer's disease, (AD), dementia with Lewy bodies (DLB) and chronic traumatic encephalopathy (CTE), now appear to be caused by the accumulation and aggregation of proteins that cause progressive damage to the brain. Recent preclinical results suggest that clearance of such neurotoxic proteins from the brain may be greatly increased during states where noradrenergic (NA) tone is decreased or blocked, such as anesthesia and normal sleep, but impaired in animal models of mild Traumatic Brain Injury (mTBI). These results also suggest that clearance through this mechanism, which has been termed the 'glymphatic' system, is likely to be decreased in conditions where NA signaling is inappropriately maintained during sleep, such as posttraumatic stress disorder (PTSD). Importantly, the rate at which toxins are cleared through the glymphatic system has been found to be under alpha-1 adrenergic receptor (AR) control, and the application of noradrenergic blockers such as the alpha-1 AR antagonist drug, prazosin, has been shown to increase waking clearance of these proteins to levels normally found during sleep or anesthesia. This suggests two important possibilities: first, that conditions in which the brain NA signaling is increased and sleep is impaired, such as posttraumatic stress disorder (PTSD) and mTBI, may predispose people to decreased clearance of neurotoxic proteins associated with the development and progression of dementia; and second, that the use of prazosin may be able to prevent such effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years of age or older
* Ability to complete psychometric and other clinical assessments in English
* No clinically significant laboratory abnormalities at screen
* Platelet count >100,000/mm2 within two weeks of lumbar puncture (LP)
* Body mass index (BMI) between 18 and 36 inclusive (BMIs outside this range affect CSF biomarker measurements and/or make LPs for CSF collection difficult to perform).
* Women of childbearing potential must agree to abstain from sexual relations that could result in pregnancy or use an effective method of birth control acceptable to both participant and the study clinician during the study. Men are not required to use contraception during the study
* Meeting criteria for at least one of the following:

  1. History of mild or moderate TBI:
* Exposure to at least one blast or experiencing at least one collision of the head associated with acute symptoms that meet VA/DoD criteria for mild or moderate TBI (loss of consciousness, if present, <24 hours; posttraumatic amnesia, if present, <1 week; Glasgow Coma Scale (if available) 9-15) ->6 months since last TBI. 2. Documented diagnosis of PTSD related to combat trauma (from any conflict)

Exclusion Criteria:

Medical

* History of severe TBI (Glasgow Coma Scale (if available) <9, loss of consciousness >24 hours, posttraumatic amnesia >1 week)
* Acute or unstable chronic medical illness, including unstable angina, recent myocardial infarction (within 6 months), congestive heart failure, preexisting hypotension (systolic <110) or orthostatic hypotension (systolic drop > 20mmHg after two minutes standing or any drop accompanied by dizziness), autoimmune disorders; insulin-dependent diabetes
* Chronic renal or hepatic failure, acute pancreatitis, Meniere's disease, benign positional vertigo, narcolepsy, or diagnosed untreated sleep apnea (sleep apnea currently being treated is not exclusionary).
* Contraindications to LP (e.g., spinal cord injury; deformity, severe disease or infection in the region of the lumbosacral spine; bleeding tendency, clotting abnormalities, use of anticoagulant medications, or platelet count <100,000/mm2); trauma or infection in the 4 weeks before LP
* Current pregnancy or lactation. Women of childbearing potential must agree to abstain from sexual relations that could result in pregnancy or use an effective method of birth control acceptable to both participant and the study clinician during the study. Men are not required to use contraception during the study.

Psychiatric/Behavioral

* Meets DSM(IV or 5, depending on what evaluative method was used in this subject) criteria for current schizophrenia, schizoaffective disorder, other specified or unspecified psychotic disorder, delirium, or any DSM cognitive disorder
* Current substance use disorder (except caffeine-related disorders, tobacco-related disorders, or cannabis intoxication) other than in remission for at least 3 months. The use of cannabis other than that meeting criteria for cannabis use disorder is not exclusionary. Use of cannabis will be documented.
* Current use of any stimulant, including prescribed stimulant medications
* Current use (within the past 1 month, ongoing, or expected during the study period) of any drugs that are illegal under Washington state law.
* Severe psychiatric instability or severe situational life crises, including evidence of being actively suicidal or homicidal, or any behavior which poses an immediate danger to participant or others.

Medications/Therapies

* Current use of prazosin or other alpha-1 antagonist or trazodone, or use of such agent within the 3 month period prior to when the baseline 2 visit would be scheduled (a 3-month washout is required due to the potential effects it may have on the biomarker measurements).
* Allergy or previous adverse reaction to prazosin or other alpha-1 antagonist
* Use of exclusionary medications in the 4 weeks prior to screening: selected CNS-acting medications; antipsychotics, anti-Parkinson's disease medications and CNS stimulants; Coumadin or other medications affecting coagulation and/or inflammation (low-dose aspirin and use of NSAIDs for pain will not be exclusionary); potent immune-modulating medications, such as hydrocortisone or methotrexate; anti-HIV medications.
* Use of avanafil (Stendra), sildenafil (Viagra), tadalafil (Cialis), and vardenafil (Levitra) will be not be permitted during the study dose titration period because of increased risk of hypotension in combination with alpha-1 blockers, but will be allowed at 1/2 the usual starting dose following dose titration
* Current use of stimulants or nitrates, or of alternative medications or supplements with stimulant properties (e.g., ephedra) or vasodilatory properties (e.g., nitrate containing supplements)
* Recent evidence based trauma- or sleep-focused psychotherapy, such as Prolonged Exposure therapy (PE), Cognitive Processing Therapy (CPT), Eye Movement Desensitization and Reprogramming (EMDR), Cognitive Behavioral Therapy for Insomnia (CBTi) or Image Rehearsal and Rescripting therapy for nightmares. These therapies must have been completed > 4 weeks before first baseline assessment visit (study visit 2).

Other

* Allergy or previous adverse reaction to prazosin or other alpha-1 antagonist
* Receiving another medication in another interventional study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murray A. Raskind, MD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nine subjects were consented to participate. Two subjects completed all baseline procedures and were randomized to study drug.
Period: Overall Study
Arm/Group | Prazosin | Placebo
Started | 1 | 1
Completed | 0 | 1
Not Completed | 1 | 0
Not completed — lumbar puncture not performed at early termination. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prazosin | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 52 [52 to 52] | 39 [39 to 39] | 45.5 [39 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in CSF Total-tau From Baseline to End of Study (pg/mL)
Description: an established biomarker of neurodegeneration in Alzheimer's disease.
Time Frame: 10 weeks
Population: The one prazosin participant did not under a lumbar puncture at the study termination visit.
Measure: Number; unit: pg/mL
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 0 | 1
pg/mL |  | 11

2. Primary Outcome: Change in p-tau181 From Baseline to End of Study (pg/mL)
Description: an established biomarker of neurodegeneration in Alzheimer's disease.
Time Frame: 10 weeks
Population: The one prazosin participant did not under a lumbar puncture at the study termination visit.
Measure: Number; unit: pg/mL
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 0 | 1
pg/mL |  | 2.3

3. Primary Outcome: Change in Amyloid Beta 42 From Baseline to End of Study (pg/mL)
Description: an established biomarker of neurodegeneration in Alzheimer's disease.
Time Frame: 10 weeks
Population: The one prazosin participant did not under a lumbar puncture at the study termination visit.
Measure: Number; unit: pg/mL
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 0 | 1
pg/mL |  | 235

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: 14 common potential adverse symptoms of prazosin were queried at every visit as well as an open ended query for other symptoms.
Arm/Group | Prazosin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prazosin (N=1) | Placebo (N=1)
adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
headache (General disorders) | 1 (2) | 0 (0)
insomnia (General disorders) | 1 (1) | 0 (0)
lack of energy (General disorders) | 1 (1) | 0 (0)
lightheadedness (General disorders) | 1 (2) | 0 (0)
nasal congestion (General disorders) | 1 (1) | 0 (0)
pain from root canal (General disorders) | 0 (0) | 1 (1)
weakness (General disorders) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
These results are not generalizable due to the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT03221751/Prot_SAP_000.pdf